CLINICAL TRIAL: NCT03713359
Title: Randomized, Controlled Clinical Trial for Measles - Rubella Combined Vaccine (MRVAC) Produced by POLYVAC by Technology Transfer From Japan (Phase III)
Brief Title: Clinical Trial for Measles - Rubella Combined Vaccine (MRVAC) Produced by POLYVAC (Phase III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center for Research and Production of Vaccines and Biologicals, Vietnam (Other Government)
Collaborators: Vietnam Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRVAC VX.2016.01
Record Dates: First submitted 2018-10-09; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Signs and Symptoms
Keywords: MRVAC vaccine, fever, rash
MeSH Terms: conditions — Signs and Symptoms; Fever; Exanthema

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized receiving either MRVAC or MR vaccine produced by Serum Institute, India, which was using in Vietnam National Expanded program on Immunization in the ratio of 2:1. The Participants will be received only 1 dose of vaccine at the age from 1 year to 45 years.
Who Masked: Participant
Masking Description: The first two volunteers will be assigned to the MRVAC group (code named A) and coded A001 and A002. The 3rd Volunteer will be assigned to the control group (code named B) and coded as B001. Volunteers arriving later will also be coded in this order until they meet enough subjects as required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial arm (MRVAC) (Active Comparator): Measles and Rubella combined vaccine (lyophilized) MRVAC produced by POLYVAC is live attenuated measles vaccine. Each vial of 10 doses of measles-rubella combined vaccine is reconstituted with 5.5 mL of water for injection. Each single dose 0.5 mL contains the following components:
  Live, attenuated strain AIK-C measles virus not less than 1000 PFU Live, attenuated strain Takahashi rubella virus not less than 1000 PFU Subcutaneous injection
  Interventions: Biological: Trial arm (MRVAC)
- Control arm (Active Comparator): Measles and Rubella combined vaccine produce by Serum Institute, India (lyophilized) is live attenuated Measles and Rubella vaccines being used in the Vietnam expanded immunization program was used as control arm.
  Subcutaneous injection
  Interventions: Biological: Control arm

INTERVENTIONS:
Biological: Trial arm (MRVAC) — Volunteers from 1-45 years old will be injected only one dose of MRVAC vaccine
  Arms: Trial arm (MRVAC)
Biological: Control arm — Volunteers from 1-45 years old will be injected only one dose of MRVAC vaccine
  Arms: Control arm

SUMMARY:
The study is conducted to evaluate the safety and Immunogenicity of Measles-Rubella combined vaccine MRVAC produced by POLYVAC (phase 3) on Vietnamese volunteers and to demonstrate non-inferiority on the immunogenicity of MRVAC in comparison to MR vaccine produced by Serum Institute, India.

DETAILED DESCRIPTION:
A phase III, Randomized, control study to compare the immunogenicity and safety of MRVAC vaccine produced by POLYVAC with MR vaccine licensed in Vietnam produced by Serum Institute, India.

1. Evaluate the safety of MRVAC produced by POLYVAC on Healthy Vietnamese volunteers from 1 - 45 years old.

   Evaluate the safety by the ratio of participants having following symptom/signs:
   * The ratio of immediate adverse events (local adverse events and systemic adverse events), within 30 minutes after vaccination.
   * The ratio of participants having local and systemic adverse events (including unexpected adverse events) occur within 28 days after vaccination.
   * The ratio of serious adverse events (SAEs) occur from day 0 to day 28 after vaccination. (SAEs).
2. Evaluate the immunogenicity of MRVAC produced by POLYVAC on the healthy volunteers from 1 - 45 years.

   * The rate of sero-conversion;
   * GMT (Geomatric mean Antibody titer) after vaccination.
3. Comparison the safety and immunogenicity between MRVAC and control vaccine.

ELIGIBILITY:
Inclusion Criteria:

* For children 1-2 years old: All subjects must meet all of the following criteria at the time of enroll to stduy:

  * Healthy children from 1 year to 2 years old.
  * Full-term birth: Pregnancy ≥ 37 weeks.
  * Weight at birth is at least 2.5kg.
  * Do not get any disease through a clinical examination and ask for medical history before taking part in the study (according to the prescribed information).
  * Have not injected Rubella vaccine or a combination vaccine containing Rubella vaccine.
  * Have not infected by Rubella before.
  * Parents or legal guardians agree to voluntarily consent to their child's participation in the study. Parent or legal guardian is provided basic information about the vaccine as well as benefits, obligations and meaning of participating in the trial. There must be a written consent form for your child to participate.
* For people from 1 year to 45 years old:

  * Do not get any disease through a clinical examination and ask for medical history before taking part in the study (according to the prescribed card).
  * Have not infected by Rubella before.
  * For people over 2 years old up to 18 years old: Parents or legal guardians agree to voluntarily consent to their child's participation in the study. Parent or legal guardian is provided basic information about the vaccine as well as benefits, obligations and meaning of participating in the trial. There must be a written consent form for your child to participate.
* For people aged 18 to 45: Completely volunteering to participate in the study after having been provided with basic information about the trial vaccine as well as the benefits, obligations and meaning of the trial participation. Must sign in the consent form to participate in the study.

Exclusion Criteria:

* Fever within 3 days before vaccination (body temperature ≥ 38 degrees Celsius) Persons with congenital malformations, neurological disorders, psychiatric disorders or families with neurological or psychiatric conditions or brain damage.
* Having abnormal immune status or being treated for immunological control; Being immunocompromised as a result of progressive disease treatment.
* Have received immunosuppressive drugs (steroid group) for more than 2 weeks before starting the vaccination.
* Allergy to any vaccine component including hypersensitivity reactions and anaphylactic shock to the antibiotics (Kanamycine and Erythromycin), egg products and gelatin.
* Family history of immunodeficiency.
* Have a history of high fever, seizures
* premature birth (<37 weeks) (applicable to children 1-2 years).
* Malnutrition level 3 or above (applicable to children 1-2 years).
* Have used of gamma globulin, blood transfusions within 3 months before vaccination or gamma glubolin in large doses or the use of immunosuppressive drugs within 6 months before vaccination
* Have used live vaccines within 27 days before vaccination; Have used other vaccines within 4 weeks before entry to study; Use of immunoglobulins or blood products within 3 months before vaccination;
* Is participating in trial other drugs or vaccines; Has an acute or chronic disease that affects the safety (including but not limited to: chronic liver disease, some kidney disease, progressive or unstable neurological disorders, diabetes and organ transplants).
* Having serious acute illness. Responsible doctor or doctor in charge of evaluation consider as unsuitable, such as having abnormal crying ...
* Having plan to go far from the study site between visits. - Being pregnant (for women aged 14 - 45 years)
* Trial subjects must satisfy selection criteria and not be subjected to exclusion criteria.

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 756 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | During 30 minutes and 28 days after only one dose vaccination
  1. Incidence rate of local adverse event (AE), systemic AE

SECONDARY OUTCOMES:
Antibody seroconversion | 42 to 56 days after only one dose vaccination .
  Positive seroconversion rates of Measles and Rubella neutralization antibody
Geo-mean antibody titer | Before vaccination and after 42 to 56 days vaccination only one dose
  Geo-mean antibody titer of both trial arm and control arm
Serious adverse event (SAE) | During 30 minutes and 28 days after vaccination only one dose
  Number of cases occur SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Dinh H. Duong, Ph.D, Principal Investigator — Epidemiology department - Vietnam Military Medical University.

IPD SHARING:
Plan to Share IPD: Undecided